CLINICAL TRIAL: NCT06290843
Title: Analysis of Body Balance Parameters in Children With Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Other Study IDs: AWFiS/2024_1_PE
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-01

CONDITIONS: Idiopathic Scoliosis
Keywords: Spinal deformity; AMTI platform; Balance; Postural stability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scoliosis: Children with idiopathic scoliosis
  Interventions: Procedure: Schroth method
- Control: Children without idiopathic scoliosis
  Interventions: Procedure: Schroth method

INTERVENTIONS:
Procedure: Schroth method — Exercises from Schoth method

SUMMARY:
The aim of the study is to compare body balance parameters assessed using the AMTI dynamometric platform in children with idiopathic scoliosis (with and without Schroth therapy) compared to control group.

DETAILED DESCRIPTION:
Assessment of balance parameters on the AMTI dynanometric platform in children with adolescent idiopathic scoliosis and healthy children in the same age group. Each person examined will have one trial measurement, followed by a 3-minute break. After the trial measurement, the actual examination will take place - 3 trials of 60 seconds each in 4 different variants: eyes open, eyes closed, single leg left lower limb eyes open, single leg right lower limb eyes open.The variants will be randomized.

Assessment of body posture using photo recordings taken with an OLYMPUS digital camera, which will be used to classify the type of scoliosis. Anthropometric points will be marked using a washable marker: cervical-thoracic junction C7-Th1, thoracic-lumbar junction Th12/L1, lumbosacral junction L5/S1, right and left anterior superior iliac spine (ASIS), right and left posterior superior iliac spine ( PSIS), the center of the right and left greater trochanters and the center of the lateral malleolus. Photo registration will be made in four positions: front, back, right side and left side. The camera is 3 m away from the subject and the height of the tripod is half the height of the body.

Analysis of spine X-ray images: Cobb angle, Schroth type of scoliosis, Bordering vertebrae, Apex vertebra, Vertebral rotation, Sagittal plane analysis

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic adolescent scoliosis aged 10-18 years, female,
* control group aged 10-18 years, female.

Exclusion Criteria:

* congenital spine defects,
* spine surgeries,
* neurological diseases,
* cardiological diseases,
* genetic diseases,
* rheumatological diseases,
* immunological diseases,
* endocrine diseases
* back pain,
* lower limb pain,
* past injuries of lower limbs or spine

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: children aged 11-18 years diagnosed with adolescent idiopathic scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Analysis of body balance on the AMTI force platform | Before and after 12-week therapy
  The measurement of center of pressure (anterior-posterior) (cm) in standing position with eyes open, eyes closed, single leg left lower limb eyes open, single leg right lower limb eyes open.
Analysis of body balance on the AMTI force platform | Before and after 12-week therapy
  Center of pressure (medial-lateral) (cm) in standing position with eyes open, eyes closed, single leg left lower limb eyes open, single leg right lower limb eyes open.
Analysis of body balance on the AMTI force platform | Directly before and after 12-week therapy
  Velocity (m/s) of center of pressure changes with eyes open, eyes closed, single leg left lower limb eyes open, single leg right lower limb eyes open.
Analysis of body balance on the AMTI force platform | Directly before and after 12-week therapy
  Sway area (cm2) of center of pressure with eyes open, eyes closed, single leg left lower limb eyes open, single leg right lower limb eyes open.
Photographic analysis of body posture | Directly before and after 12-week therapy
  The photos will be taken in various positions: front, back and both sides.
Analysis of x-ray in the frontal plane | One-time examintation before therapy
  Cobb angle (degree)
Analysis of x-ray in the frontal plane | One-time examintation before therapy
  Bordering vertebrae (no.)
Analysis of x-ray in the frontal plane | One-time examintation before therapy
  Apex vertebra (no.)
Analysis of x-ray in the frontal plane | One-time examintation before therapy
  Vertebral rotation (degree)
Analysis of x-ray in the sagittal plane | One-time examintation before therapy
  Kyphosis angle (degree)
Analysis of x-ray in the sagittal plane | One-time examintation before therapy
  Lordosis angle (degree)

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Ewertowska, Principal Investigator — Akademia Wychowania Fizycznego i Sportu w Gdańsku
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland